CLINICAL TRIAL: NCT03063424
Title: Hyperventilation Versus Exercise Testing Sensitivity in Exercise Induced Asthma
Acronym: HYVES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Brian Grondin-Beaudoin, Clinical Professor, Principal Investigator, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 10-074
Record Dates: First submitted 2017-01-22; First posted 2017-02-24 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Exercise Induced Bronchospasm
Keywords: isocapnic voluntary hyperventilation; eucapnic voluntary hyperventilation; exercise induced bronchoconstriction; exercise challenge cycle ergometer
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Other)
  Interventions: Diagnostic Test: Eucapnic voluntary hyperventilation; Diagnostic Test: Exercise challenge on a cycle ergometer
- Asthmatics with EIB (Other)
  Interventions: Diagnostic Test: Eucapnic voluntary hyperventilation; Diagnostic Test: Exercise challenge on a cycle ergometer

INTERVENTIONS:
Diagnostic Test: Eucapnic voluntary hyperventilation
Diagnostic Test: Exercise challenge on a cycle ergometer

SUMMARY:
The diagnosis of exercise-induced bronchospasm (EIB) is difficult. The metacholine challenge test is not enough specific for the diagnosis of EIB. The exercise challenge test on a cycle ergometer is often use to diagnose this condition. This test has very high specificity, but not enough sensibility because the ventilation achieved during this test is often not big enough to induce a bronchospasm, especially in trained athletes. Eucapnic voluntary hyperventilation (EVH) is the recommended test of the Olympic National committee to establish the diagnosis of EIB, but there are no study comparing the sensibility and specificity of the cycle ergometer challenge test and the isocapnic hyperventilation in an establish population of asthmatics. The investigators assume that the sensitivity and specificity of EVH are higher than those of the cycle ergometer for the diagnosis of EIB in a population of asthmatics with symptoms suggestive of bronchospasm on exertion. In a population of asthmatics with exercise symptoms, what is the sensitivity and specificity of EVH and exercise challenge on a cycle ergometer for the diagnosis of EIB?

ELIGIBILITY:
Inclusion Criteria for the group "exercise-induced bronchospasm":

* The subject must have a diagnosis of asthma according to 2010 Canadian Thoracic Society consensus criteria since more then one year.
* The subject should have an average expiratory volume per second (FEV1) ≥ 80% of the predicted value (post bronchodilatation) at the time of the initial visit.
* The subject must have had a positive methacholine test at the first visit of the study demonstrating the presence of bronchial hyperreactivity.
* The subject must have asthma control as defined by 2010 Canadian Thoracic Society consensus, with the obvious exception of limitations related to physical activity.
* The subject must have at the questionnaire significant symptoms of exercise-induced bronchospasm for more than 6 months.

Inclusion Criteria for the group "healthy":

* The subject should not have a positive history of eczema, urticaria or allergic rhinitis for life.
* The subject should have a FEV1 ≥ 80% of the predicted value and an FEV1 / FVC (Forced vital capacity) ratio of ≥70% at the time of the initial visit.
* The subject should have a negative methacholine test at the first visit of the study.
* The subject should not exhibit symptoms considered clinically compatible with EIB diagnosis.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* The subject should not suffer from clinically significant concomitant diseases that may compromise the course of the study.
* The subject should not have taken per os or intravenously steroids in the 8 weeks prior to the study.
* The subject should not have experienced significant symptoms of respiratory tract infection (viral or bacterial) in the 8 weeks prior to the study.
* The subject must not have participated in another study during the month preceding the date of enrollment of this study.
* The subject should not have smoked within the last 6 months.

Exclusion criteria during the study:

* The subject doesn't show up for all 3 visits or doesn't complete all required exams.
* The subject develops a respiratory tract infection, an acute exacerbation of his asthma or any other conditions that compromise his participation in the required examinations.
* The subject has a pre-test FEV1 of less than 80%.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Compare the sensitivity and specificity of eucapnic voluntary hyperventilation versus exercise challenge testing on a cycle ergometer for exercise-induced bronchospasm diagnosis in established asthmatic subjects with exercise symptoms. | through study completion, an average of 1 month

SECONDARY OUTCOMES:
Correlate the magnitude of exercise bronchoconstriction during EVH and exercise challenge testing on a cycle ergometer (measurement of FEV1 before and after these tests) with severity of symptoms of EIB (with questionnaires) | through study completion, an average of 1 month
  The questionnaires for the severity of symptoms of EIB will include a modified Borg questionnaire, symptoms of EIB after the tests and usual symptoms of EIB after a vigorous effort.
Correlate the magnitude of exercise bronchoconstriction during EVH and exercise challenge testing on a cycle ergometer (FEV1 before and after these tests) with severity of bronchial hyperreactivity evaluated by methacholine challenge test (MCT). | through study completion, an average of 1 month
  severity of bronchial hyperreactivity evaluated by methacholine challenge test (MCT) will be measured with the provocative concentration causing a 20% fall in FEV1 (PC20) (mg/ml) as recommended by the American Thoracic Society (ATS).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Larivée, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided